CLINICAL TRIAL: NCT03944538
Title: Physical Activity Intervention for Improving Vascular Comorbidity Risk in Multiple Sclerosis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Research restrictions and recruitment challenges due to the COVID-19 pandemic
Sponsor: University of Ottawa (Other)
Collaborators: University of Illinois at Chicago (Other); National Multiple Sclerosis Society (Other)
Responsible Party: Principal Investigator, Lara Pilutti, Associate Professor, University of Ottawa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: H09-17-06
Record Dates: First submitted 2019-05-06; First posted 2019-05-09 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2023-05

CONDITIONS: Multiple Sclerosis
Keywords: Exercise; Fitness; Co-morbidity
MeSH Terms: conditions — Multiple Sclerosis; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lifestyle Physical Activity (Experimental): The primary content of the website will be delivered through interactive video courses. The courses will be released seven times during the first two months, four times during the second two months, and twice during the final two months of the intervention.
  The website Tracker feature will allow for tracking of daily step counts as well as setting goals and monitoring progress.
  The one-on-one video chats will be conducted face to face through Zoom and will be semi-scripted. The chats will consist of an ongoing review of goal-setting and progress toward goal attainment through Tracker as well as discussion of strategies and facilitators of behavioral changes based on social cognitive theory and current website content. The chats will occur at the same frequency as the video course release. For the second 6 months of the study, participants will be asked to maintain their usual activities.
  Interventions: Behavioral: Lifestyle Physical Activity
- General Wellness (Active Comparator): The general wellness condition will focus on self-managing MS through means other than physical activity. The materials are transformations of brochures provided by the National Multiple Sclerosis Society. The delivery of the Internet materials and chat sessions will occur on the same schedule and frequency as the intervention condition, and will have a comparable time commitment. This condition will account for attention and social contact as well as other possible biases such as initial reactivity and time spent on the website and video chats. For the second 6 months of the study, participants will be asked to maintain their usual activities.
  Interventions: Behavioral: General Wellness

INTERVENTIONS:
Behavioral: Lifestyle Physical Activity — The intervention consists of two primary components: a dedicated Internet website and one-on-one video chats with a behavioral coach via Zoom. The intervention focuses on the skills, techniques, resources and strategies for becoming and staying physically active with MS, but does not provide a prescription for exercise or physical activity itself.
  Arms: Lifestyle Physical Activity
Behavioral: General Wellness — The control condition provides an Internet website and one-on-one video chats that discuss materials about self-managing MS consequences and health indicators through methods other than physical activity.
  Arms: General Wellness

SUMMARY:
Vascular comorbidities, such as high cholesterol, obesity, high blood pressure, and diabetes, are common among people with multiple sclerosis (MS), and can negatively impact disease diagnosis, treatment, and progression. Physical inactivity may be one possible reason for this increased risk and may occur through changes in cardiorespiratory fitness (the ability of the body to transport and use oxygen during sustained physical activity). While exercise training is effective for improving fitness, factors such as accessibility to facilities and financial cost may not make it a viable option for most people with MS. An alternative approach for improving fitness is by increasing daily physical activity levels. The research team has developed and tested an Internet-delivered lifestyle physical activity intervention that has been shown to improve physical activity levels among people with MS. This lifestyle intervention is a promising approach for also increasing fitness and managing vascular comorbidity risk in persons with MS. This randomized clinical trial will examine the efficacy of a 6-month lifestyle physical activity intervention on cardiorespiratory fitness and vascular comorbidity risk in persons with MS.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of multiple sclerosis
* Relapse-free in the past 30 days
* Stable course of disease modifying therapy over the past 6 months
* Being non-active, defined as not engaging in regular exercise (i.e., ≥30 minutes/day on >2 days/week during the last 6 months)
* Internet access
* Ability to comprehend study materials and communicate in English
* Expanded Disability Status Scale (EDSS) score <6.0
* Willingness to complete three testing sessions at the University of Ottawa separated by 6 months
* Willing to undergo randomization to a lifestyle physical activity condition or general wellness condition for 6 months
* Intermediate risk level for cardiovascular disease based on the Framingham Cardiovascular Disease Risk Score calculator
* Asymptomatic (i.e., no major signs or symptoms of acute or uncontrolled cardiovascular, metabolic, or renal disease; e.g., chest pain) based on the Get Active Questionnaire and the health history section of the American Heart Association (AHA)/American College of Sports Medicine (ACSM) Health/Fitness Facility Pre-participation Screening Questionnaire
* Physician approval for participation

Exclusion Criteria:

* Pregnancy
* Previous enrollment in lifestyle physical activity behaviour interventions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2019-07-21 (Actual); Primary Completion 2020-10-20 (Actual); Study Completion 2020-10-20 (Actual)

PRIMARY OUTCOMES:
Change in Cardiorespiratory Fitness | Change in cardiorespiratory fitness from baseline at 6- and 12-months
  Peak oxygen consumption (VO2peak) measured using an incremental exercise test and metabolic measurement system for analyzing expired gases

SECONDARY OUTCOMES:
Change in Blood Pressure | Change in blood pressure from baseline at 6- and 12-months
  Systolic and diastolic blood pressure following 5-10 min rest
Change in Body Composition | Change in body composition from baseline at 6- and 12-months
  Fat and lean soft tissue masses assessed using dual-energy X-ray absorptiometry
Change in Blood Glucose | Change in blood glucose from baseline at 6- and 12-months
  Fasting blood glucose measured in venous blood
Change in Insulin Resistance | Change in insulin resistance from baseline at 6- and 12-months
  Homeostatic Model Assessment of insulin resistance (HOMA-IR)
Change in Triglycerides and Cholesterols | Change in triglycerides and cholesterols from baseline at 6- and 12-months
  Fasting blood triglycerides and cholesterols (total cholesterol, high-density lipoprotein cholesterol, low-density lipoprotein cholesterol) measured in venous blood

OTHER OUTCOMES:
Neurological Function - Expanded Disability Status Scale | Baseline, 6-months and 12-months
  The Expanded Disability Status Scale is a standard neurological examination for persons with MS. The scale is used to assess neurological function within eight functional systems: pyramidal, cerebellar, brainstem, sensory, bowel and bladder, visual, cerebral, and other. The total score generated for each participant ranges between 0 (normal neurological function) to 10 (death due to MS).
Dietary Intake | Baseline, 6-months and 12-months
  3-day diet log
Change in Physical Activity - assessed by accelerometry | Change in physical activity from baseline at 6- and 12-months
  Minutes per day of moderate-to-vigorous and light physical activity, and sedentary time
Change in Physical Activity - assessed by Godin Leisure-Time Exercise Questionnaire | Change in physical activity from baseline at 6- and 12-months
  The Godin Leisure-Time Exercise Questionnaire includes three items that measure the frequency of vigorous, moderate, and light physical activities that occur for at least 15 minutes during one's leisure-time over the previous 7 days. The three items are weighted and then summed into a total score that can range between 0 (low active) to 119 (high active).
Change in Body Circumferences | Change in body circumferences from baseline at 6- and 12-months
  Waist and hip circumferences
Change in Optical Coherence Tomography (OCT) measures | Change in OCT measures from baseline at 6- and 12-months
  Retinal nerve fibre layer thickness will be assessed using OCT

CONTACTS AND LOCATIONS:
Overall Officials: Lara Pilutti, PhD, Principal Investigator — University of Ottawa
Locations (1):
- University of Ottawa, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Platta ME, Ensari I, Motl RW, Pilutti LA. Effect of Exercise Training on Fitness in Multiple Sclerosis: A Meta-Analysis. Arch Phys Med Rehabil. 2016 Sep;97(9):1564-1572. doi: 10.1016/j.apmr.2016.01.023. Epub 2016 Feb 16. PMID 26896750
- [Background] Motl RW, Goldman M. Physical inactivity, neurological disability, and cardiorespiratory fitness in multiple sclerosis. Acta Neurol Scand. 2011 Feb;123(2):98-104. doi: 10.1111/j.1600-0404.2010.01361.x. PMID 21108624
- [Background] Pilutti LA, Dlugonski D, Sandroff BM, Klaren R, Motl RW. Randomized controlled trial of a behavioral intervention targeting symptoms and physical activity in multiple sclerosis. Mult Scler. 2014 Apr;20(5):594-601. doi: 10.1177/1352458513503391. Epub 2013 Sep 5. PMID 24009162
- [Background] Pilutti LA, Dlugonski D, Sandroff BM, Klaren RE, Motl RW. Internet-delivered lifestyle physical activity intervention improves body composition in multiple sclerosis: preliminary evidence from a randomized controlled trial. Arch Phys Med Rehabil. 2014 Jul;95(7):1283-8. doi: 10.1016/j.apmr.2014.03.015. Epub 2014 Mar 31. PMID 24699237